CLINICAL TRIAL: NCT04516798
Title: The Reflex Mechanism Underlying The Neuromuscular Effects Of The Whole Body Vibration
Brief Title: The Reflex Mechanism Underlying Neuromuscular Effects Of The Whole Body Vibration
Acronym: WBV-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ISTANBULPMR
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Reflex, Ankle, Decreased
Keywords: whole body vibration; tonic vibration reflex; muscle spindle
MeSH Terms: conditions — Reflex, Abnormal | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: Self controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): Local and whole body vibration were applied
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — local and whole-body vibration were applied

SUMMARY:
This study was conducted to determine whether the spinal reflex mechanism underlying the neuromuscular effects of whole body vibration (WBV) is tonic vibration reflex. Local and whole body vibration reflex latencies were measured in young adult healthy volunteers.

DETAILED DESCRIPTION:
A total of eight volunteers were included according to the inclusion and exclusion criteria. The subjects were vibrated while standing upright with the WBV device (PowerPlate® Pro5). The 30, 35 and 40 Hz WBVs were applied for thirty seconds for each frequency with an amplitude of 2 mm. In the same session, 100, 135 and 150 Hz local vibrations were applied to the right Achilles tendon for thirty seconds for each frequency. 100, 135 and 150 Hz local vibrations were then applied to the right heel for thirty seconds for each frequency with an interval of five seconds. Vibration stimuli were recorded accelerometers. Reflex muscle responses were recorded from the right soleus muscle at a sampling rate of 40 KHz. Recording electrodes were placed on the belly of the right soleus muscle and the ground electrode was placed on the right medial malleolus.

The data were recorded with the PowerLab device, the records were processed and analyzed offline from the LabChart program. After the EMG records are filtered and rectified, reflex latencies were measured by cumulative averaging method using the accelerometer records as triggers (Karacan I, Cakar HI, Sebik O, Yilmaz G, Cidem M, Kara S, Türker KS.A new method to determine reflex latency induced by high rate stimulation of the nervous system.Front Hum Neurosci.2014 Jul 18; 8: 536.doi: 10.3389 / fnhum.2014.00536). After determining the Achilles tendon vibration reflex latency and the reflex latency induced by WBV, it was compared with statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Young adult (20-40 years old)
* Both gender
* Volunteer

Exclusion Criteria:

* Cardiac disorder (Rhythm / conduction disorder, Cardiac pacemaker, Ischemic heart disease)
* Finding or suspected active deep vein thrombosis,
* History of deep vein thrombosis and pulmonary embolism,
* Orthostatic hypotension
* Hypertension
* Presence of fracture in the lower limb
* Achilles Contractures
* Active inflammatory, rheumatological or infectious disease in the lower limb
* Peripheral nerve lesions such as polyneuropathy, radiculopathy in the lower limb
* Those with a history of Achilles tendinopathy / bursitis
* Those with a history of kidney stones
* Patients with dizziness and balance problems,
* Cases with lesions on the skin surface where electrodes were attached
* Those with communication-cooperation problems
* Having a history of panic attacks

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
reflex latency | during intervention, an average of 8 minutes
  The time between the vibration stimulus and the reflex muscle response triggered by it was defined as the latency.

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan Karacan, Assoc Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildirim MA, Topkara B, Aydin T, Paker N, Soy D, Coskun E, Ones K, Bardak A, Kesiktas N, Ozyurt MG, Celik B, Onder B, Kilic A, Kucuk HC, Karacan I, Turker KS. Exploring the receptor origin of vibration-induced reflexes. Spinal Cord. 2020 Jun;58(6):716-723. doi: 10.1038/s41393-020-0419-5. Epub 2020 Jan 15. PMID 31942042
- [Result] Aydin T, Kesiktas FN, Baskent A, Karan A, Karacan I, Turker KS. Cross-training effect of chronic whole-body vibration exercise: a randomized controlled study. Somatosens Mot Res. 2020 Jun;37(2):51-58. doi: 10.1080/08990220.2020.1720635. Epub 2020 Feb 5. PMID 32024411
- [Result] Karacan I, Cakar HI, Sebik O, Yilmaz G, Cidem M, Kara S, Turker KS. A new method to determine reflex latency induced by high rate stimulation of the nervous system. Front Hum Neurosci. 2014 Jul 18;8:536. doi: 10.3389/fnhum.2014.00536. eCollection 2014. PMID 25100978